CLINICAL TRIAL: NCT06846866
Title: A Phase 1, Double-blind, Placebo-controlled, Randomized Study of the Safety, Tolerability, and Pharmacokinetics of BMS-986419 (Part 1) and a Phase 1 Randomized, Double-blind, Positive-controlled, Placebo-controlled, Parallel, Nested-crossover (Moxifloxacin-placebo) Thorough QT/QTc Study to Evaluate the Effect of Multiple Doses of BMS-986419 on Cardiac Repolarization (Part 2) in Healthy Participants
Brief Title: A Study to Investigate the Safety, Tolerability, and Drug Levels of BMS-986419 (Part 1) and the Effects Multiple Doses of BMS-986419 on Cardiac Repolarization (Part 2) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CN007-1005
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers
Keywords: BMS-986419, healthy, QTC, pharmacokinetics, moxifloxacin
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: Administration of BMS-986419 (Experimental)
  Interventions: Drug: BMS-986419
- Part 1: Administration of Placebo (Placebo Comparator)
  Interventions: Drug: BMS-986419 Matching Placebo
- Part 2: Group 1 (Experimental)
  Interventions: Drug: BMS-986419; Drug: BMS-986419 Matching Placebo; Drug: Moxifloxacin Matching Placebo
- Part 2: Group 2a (Experimental)
  Interventions: Drug: BMS-986419 Matching Placebo; Drug: Moxifloxacin; Drug: Moxifloxacin Matching Placebo
- Part 2: Group 2b (Experimental)
  Interventions: Drug: BMS-986419 Matching Placebo; Drug: Moxifloxacin; Drug: Moxifloxacin Matching Placebo

INTERVENTIONS:
Drug: BMS-986419 — Specified dose on specified days
  Arms: Part 1: Administration of BMS-986419; Part 2: Group 1
Drug: BMS-986419 Matching Placebo — Specified dose on specified days
  Arms: Part 1: Administration of Placebo; Part 2: Group 1; Part 2: Group 2a; Part 2: Group 2b
Drug: Moxifloxacin — Specified dose on specified days
  Arms: Part 2: Group 2a; Part 2: Group 2b
Drug: Moxifloxacin Matching Placebo — Specified dose on specified days
  Arms: Part 2: Group 1; Part 2: Group 2a; Part 2: Group 2b

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, and pharmacokinetics of BMS-986419 (Part 1) and the effects of multiple doses of BMS-986419 on cardiac repolarization (Part 2) in healthy participants.

ELIGIBILITY:
Inclusion Criteria

* Participants must be healthy as determined by medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory assessments.
* Participants must have a Body mass index (BMI) between 18.0 and 30.0 kilograms/meter square (kg/m^2), inclusive, at screening.

Exclusion Criteria

* Participants must not have any significant acute or chronic medical illness as determined by the investigator.
* Participants must not have any current or recent (within 3 months of study intervention administration) GI disease, liver and kidney that could possibly affect drug absorption, distribution, metabolism, and excretion, (e.g., bariatric procedure, Cholecystectomy, and any other GI surgery that could impact upon the absorption of study intervention).
* Participants must not have Gilbert Syndrome.
* Participants must not have a history of clinically relevant cardiac disease as determined by the investigator, symptomatic or asymptomatic arrhythmias, presyncope or syncopal episodes, or additional risk factors for ventricular arrhythmias (e.g., long QT syndrome, catecholamine polymorphic ventricular tachycardia).
* Participants must not have exposure to any investigational drug or placebo (other than BMS-986419 or moxifloxacin) within 4 weeks or 5 half-lives (whichever is longer) prior to Day -1 (Day -2 for Part 2) until follow-up phone call.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Non-serious Adverse Events (NSAEs) | Up to approximately Day 42
Part 1: Number of Participants with Serious Adverse Events (SAEs) | Up to approximately Day 42
Part 1: Number of Participants with AEs Leading to Discontinuation | Up to approximately Day 42
Part 1: Number of Participants With AEs of Special Interest (AESI) | Up to approximately Day 42
Part 1: Number of Participants With Clinically Significant Vital Sign Abnormalities | Up to approximately Day 21
  Vital sign parameters include temperature, systolic blood pressure (BP), diastolic BP, respiratory rate, and heart rate (HR) assessment.
Part 1: Number of Participants With Clinically Significant Laboratory Assessment Abnormalities | Up to approximately Day 21
Part 1: Number of Participants With Clinically Significant 12-Lead Electrocardiogram (ECG) Abnormalities | Up to approximately Day 21
Part 1: Number of Participants With Clinically Significant Columbia-Suicide Severity Rating Scale (C-SSRS) Abnormalities | Up to approximately Day 21
Part 1: Number of Participants With Clinically Significant Neurological Examination Abnormalities | Up to approximately Day 21
Part 1: Number of Participants With Physical Examination Abnormalities | Up to approximately Day 21
Part 2: ΔQTc: Change From Baseline in Plasma Concentration of BMS-986419 on Cardiac Repolarization Expressed by QT interval (QTc) | Up to approximately Day 15
  ΔQTc is performed by primary correction.
Part 2: ΔΔQTc: Placebo-corrected Change From Baseline QTc Plasma Concentration of BMS-986419 on Cardiac Repolarization Expressed by QTc | Up to approximately Day 15

SECONDARY OUTCOMES:
Part 1: Maximum Observed Plasma Concentration (Cmax) of BMS-986419 | Up to approximately Day 21
Part 1: Time of Maximum Plasma Observed Concentration (Tmax) of BMS-986419 | Up to approximately Day 21
Part 1: Area Under the Concentration-time Curve in One Dosing Interval (AUC(TAU)) of BMS-986419 | Up to approximately Day 21
Part 1: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC [0-T]) of BMS-986419 | Up to approximately Day 21
Part 1: Terminal Phase Elimination Half-life (T-Half) of BMS-986419 | Up to approximately Day 21
Part 1: Accumulation Index; Ratio of Cmax at Steady-state to Cmax After the First Dose (AI_Cmax) of BMS-986419 | Up to approximately Day 21
Part 1: Accumulation Index; Ratio of AUC(TAU) at Steady-state to AUC(TAU) After the First Dose [AI_AUC(TAU)] of BMS-986419 | Up to approximately Day 21
Part 1: Apparent Total Body Clearance (CLT/F) of BMS-986419 | Up to approximately Day 21
Part 1: Apparent Volume of Distribution of Terminal Phase (Vz/F) of BMS-986419 | Up to approximately Day 21
Part 1: Trough Concentration of BMS-986419 | Up to approximately Day 21
Part 2: ΔQTc of BMS-986419 Using Change From Baseline of Heart Rate (HR)(ΔHR) Correction | Up to approximately Day 15
Part 2: ΔQTc of BMS-986419 Using Change From Baseline of Pulse Rate (PR)(ΔPR) Correction | Up to approximately Day 15
Part 2: ΔQTc of BMS-986419 Using Change From Baseline of Respiratory Rate (RR) Interval Correction | Up to approximately Day 15
Part 2: Change From Baseline of BMS-986419 in Quality Rating System (QRS) Interval (ΔQRS) | Up to approximately Day 15
Part 2: Number of Participants With Treatment-emergent Values of Fridericia's Corrected QT interval (QTcF) for BMS-986419 | Up to approximately Day 15
  Participants with increase in absolute treatment-emergent QTc values >450 and ≤480 milliseconds (msec), >480 and ≤500 msec, or >500 msec, and changes from pre-dose baseline of >30 and ≤ 60 msec, or >60 msec will be measured.
Part 2: Number of Timepoints With Change in Absolute Treatment-emergent QTcF Values for BMS-986419 | Up to approximately Day 15
  Number of timepoints with increase in absolute treatment-emergent QTc values >450 and ≤480 milliseconds (msec), >480 and ≤500 msec, or >500 msec, and changes from pre-dose baseline of >30 and ≤ 60 msec, or >60 msec will be measured.
Part 2: Number of Participants With Treatment-emergent Values of Individualized Heart Rate-corrected Interval/Optimized HR-corrected QT Interval (QTcS/QTcI) for BMS-986419 | Up to approximately Day 15
Part 2: Number of Participants With Treatment-emergent Values of HR for BMS-986419 | Up to approximately Day 15
  Participants with decrease in HR from pre-dose baseline >25% to a HR <50 beats per minute (bpm); and increase in HR from pre-dose baseline >25% to a HR >100 bpm will be determined.
Part 2: Number of Timepoints With Change in Absolute Treatment-emergent HR Values for BMS-986419 | Up to approximately Day 15
  Number of timepoints with decrease in HR from pre-dose baseline >25% to a HR <50 beats per minute (bpm); and increase in HR from pre-dose baseline >25% to a HR >100 bpm will be determined.
Part 2: Number of Participants With Treatment-emergent Values of PR for BMS-986419 | Up to approximately Day 15
  Participants with increase in PR from pre-dose baseline >25% to a PR>200 msec will be determined.
Part 2: Number of Timepoints With Increase in Absolute Treatment-emergent PR Values for BMS-986419 | Up to approximately Day 15
  Number of timepoints with increase in PR from pre-dose baseline >25% to a PR>200 msec will be determined.
Part 2: Number of Participants With Treatment-emergent Values of QRS for BMS-986419 | Up to approximately Day 15
  Participants with increase in QRS from pre-dose baseline >25% to a QRS >120 msec will be determined.
Part 2: Number of Timepoints With Increase in Absolute Treatment-emergent QRS Values for BMS-986419 | Up to approximately Day 15
  Number of timepoints with increase in QRS from pre-dose baseline >25% to a QRS >120 msec will be determined.
Part 2: Number of Participants With New Onset ECG Morphology Findings | Up to approximately Day 15
  "New" means an ECG finding that is not present on any baseline ECG [that is, any ECG recorded prior to receipt of the first dose of study BMS-986419] and becomes present on at least 1 on-treatment ECG during that treatment period).
Part 2: ΔQTc: Change From Baseline in Plasma Concentration of Moxifloxacin on Cardiac Repolarization Expressed by QT interval (QTc) | Up to approximately Day 15
  ΔQTc is performed by primary correction.
Part 2: ΔΔQTc: Placebo-corrected Change From Baseline QTc Plasma Concentration of Moxifloxacin on Cardiac Repolarization Expressed by QTc | Up to approximately Day 15
Part 2: Number of Participants with NSAEs | Up to approximately Day 36
Part 2: Number of Participants with SAEs | Up to approximately Day 36
Part 2: Number of Participants with AEs Leading to Discontinuation | Up to approximately Day 36
Part 2: Number of Participants With AESI | Up to approximately Day 36
Part 2: Number of Participants With Clinically Significant Vital Sign Abnormalities | Up to approximately Day 15
  Vital sign parameters include temperature, systolic BP, diastolic BP, respiratory rate, and HR assessment.
Part 2: Number of Participants With Clinically Significant Laboratory Assessment Abnormalities | Up to approximately Day 14
Part 2: Number of Participants With Clinically Significant 12-Lead ECG Abnormalities | Up to approximately Day 15
Part 2: Number of Participants With Clinically Significant C-SSRS Abnormalities | Up to approximately Day 15
Part 2: Number of Participants With Clinically Significant Neurological Examination Abnormalities | Up to approximately Day 15
Part 2: Number of Participants With Physical Examination Abnormalities | Up to approximately Day 15
Part 2: Cmax of BMS-986419 | Up to approximately Day 15
Part 2: Tmax of BMS-986419 | Up to approximately Day 15
Part 2: AUC(0-T) of BMS-986419 | Up to approximately Day 15
Part 2: AUC(TAU) of BMS-986419 | Up to approximately Day 15
Part 2: T-Half of BMS-986419 | Up to approximately Day 15
Part 2: AI_Cmax of BMS-986419 | Up to approximately Day 15
Part 2: AI_AUC(TAU) of BMS-986419 | Up to approximately Day 15
Part 2: Trough Concentration of BMS-986419 | Up to approximately Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com